CLINICAL TRIAL: NCT05849779
Title: Randomized Clinical Trial of Inhaled Sedation With Sevoflurane in Critically Ill Patients at Risk of Developing the Acute Respiratory Distress Syndrome
Brief Title: Inhaled Sevoflurane for ARDS Prevention
Acronym: IPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPA trial (AOI 2019 JABAUDON)
Record Dates: First submitted 2023-04-27; First posted 2023-05-09 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Sedation; Inhaled sevoflurane
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, single-center, prospective, randomized, stratified, parallel-group clinical trial with blinded outcome assessment and concealed allocation of patients at risk of developing the ARDS to a strategy of inhaled sedation with sevoflurane or to a strategy of current intravenous sedation practice.
Who Masked: Outcomes Assessor
Masking Description: Patients will be followed up for primary and secondary endpoints by members of the research staff who will be unaware of the trial group allocation. Information on whether the primary and secondary outcomes occur will be collected and entered into the electronic web-based case report form (eCRF) by trial or clinical trained personal (clinical research associate), blinded to the allocation group, under the supervision of the local principal investigator (PI) or designee who will also be unaware of the trial group allocation.
  Finally, the independent trial statistician and the members of the data monitoring and safety committee (DMSC) will also remain blinded for the allocation during analysis. However, the observation of differences in serious adverse events between the two groups will allow, for safety reasons may the DMSC deem necessary, to unblind allocation groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled sedation with sevoflurane (Experimental): Sevoflurane as vaporized via the Anesthesia Conserving Device (Sedaconda-ACD-S, Sedana Medical, Danderyd, Sweden).
  Interventions: Drug: Inhaled sedation with sevoflurane
- Intravenous sedation (Active Comparator): The investigators will not mandate the sedative type, but rather encourage the use of sedatives that are already routinely used in participating ICUs (typically a benzodiazepine, propofol, or dexmedetomidine, i.e. drugs approved for sedation).
  Interventions: Drug: Intravenous sedation (current practice)

INTERVENTIONS:
Drug: Inhaled sedation with sevoflurane — In both arms, the management of sedation will be conducted in the broader picture of ICU patient care, as per current standard practice in participating ICUs, and following the current guidelines for Pain, Agitation, Delirium, Immobility, and Sleep Disruption (PADIS) published in 2018 by the Society of Critical Care Medicine.
  Among many recommendations, this will include the monitoring and titration of both sedation and analgesia using validated scores such as the Richmond Agitation-Sedation Scale (RASS) for sedation. As a result of the current recommendations, the level, dose, and duration of sedation will vary among patients and will be decided by the treating clinicians. The choice of the analgesic drug(s) will be as per the treating clinicians.
  Other aspects of critical care will adhere to standard care, including the use of the "Checklist for Lung Injury Prevention" (CLIP).
  Other Names: Experimental
  Arms: Inhaled sedation with sevoflurane
Drug: Intravenous sedation (current practice) — In both arms, the management of sedation will be conducted in the broader picture of ICU patient care, as per current standard practice in participating ICUs, and following the current guidelines for Pain, Agitation, Delirium, Immobility, and Sleep Disruption (PADIS) published in 2018 by the Society of Critical Care Medicine.
  Among many recommendations, this will include the monitoring and titration of both sedation and analgesia using validated scores such as the Richmond Agitation-Sedation Scale (RASS) for sedation. As a result of the current recommendations, the level, dose, and duration of sedation will vary among patients and will be decided by the treating clinicians. The choice of the analgesic drug(s) will be as per the treating clinicians.
  Other aspects of critical care will adhere to standard care, including the use of the "Checklist for Lung Injury Prevention" (CLIP).
  Other Names: Control
  Arms: Intravenous sedation

SUMMARY:
This study focuses on patients who are at risk of developing a serious, life-threatening respiratory disease called Acute Respiratory Distress Syndrome (ARDS), which severely disrupts the function of their lungs.

Preclinical studies have shown that the use of a volatile anesthetic agent such as Sevoflurane could be beneficial in the treatment and prevention of this respiratory condition. By improving gas exchange and attenuating pulmonary inflammation in particular, this agent would make it possible to prevent deterioration or to restore pulmonary function more rapidly.

Half of the patients will receive inhaled sedation with sevoflurane and the other half will receive intravenous sedation already routinely used in participating ICUs (typically propofol, dexmedetomidine or a benzodiazepine, i.e. drugs approved for sedation).

The aim of this study is to assess whether the use of Sevoflurane could be beneficial in the prevention of ARDS.

DETAILED DESCRIPTION:
MAIN OBJECTIVE To assess the efficacy of inhaled sevoflurane, compared to current intravenous sedation practice, for improving PaO2/FiO2 in ICU patients at high risk for ARDS.

HYPOTHESIS The investigators hypothesized that a strategy of inhaled sedation with sevoflurane could be more effective than current intravenous sedation practice at improving pulmonary function during the early days of ICU admission, in patients at risk of ARDS.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to participating ICUs with at least one known risk factor for ARDS and a LIPS equals to, or greater than, 4 (Appendix D)105
3. Patient under invasive mechanical ventilation
4. With expected duration of sedation superior or equal to 4 hours
5. Affiliation to the French Sécurité Sociale

Exclusion Criteria:

* Patient under judicial protection, guardianship or supervision, as defined by art L1121-8 of the Public Health Code
* Patient under psychiatric care as defined by art. L1121-6 of the Public Health Code
* Patient deprived of their freedom by judiciary or administrative order
* Known pregnancy
* Presence of ARDS prior to randomization
* Endotracheal ventilation for greater than 24 hours prior to randomization
* Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BIPAP used solely for sleep-disordered breathing
* Tidal volume of 6 mL/kg predicted body weight (PBW) below 200 mL (i.e. height inferior to 134cm for a man and 139cm for a woman)
* Moribund patient, i.e. not expected to survive 24 hours despite intensive care
* Previous hypersensitivity or anaphylactic reaction to sevoflurane or to the intravenous sedation agent routinely used in the participating ICU (such as midazolam, propofol, or dexmedetomidine)
* Absolute contra-indications to the intravenous sedation agent routinely used in the participating ICU (such as midazolam, propofol, or dexmedetomidine)
* Medical history of malignant hyperthermia
* Long QT syndrome at risk of arrhythmic events
* Medical history of liver disease attributed to previous exposure to a halogenated agent (including sevoflurane)
* Suspected or proven intracranial hypertension
* Enrollment in another interventional trial with direct impact on oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | within 5 days from randomization
  longitudinal evolution in the PaO2/FiO2 ratio

SECONDARY OUTCOMES:
Progression to ARDS | within 5 days from randomization
  Progression to ARDS will be assessed according to the Berlin criteria, including chest radiographs
Rate of pneumonia | Presence of pneumonia will be assessed daily until Day 5, and at Day 28 or ICU discharge, whichever comes first.
  Pneumonia will be defined according to the 3 following criteria:
  * Two chest radiographs showing signs of pneumonia, or one in absence of cardiomyopathy or underlying pulmonary condition.
  * One item among: body temperature ≥38.3°C without evident cause, leukocytes <4000/mm3 or ≥12000/mm3
  * Two items among: purulent secretions, cough or dyspnea, increased need for oxygen supplementation or ventilatory assistance.
Ventilator-free days to day 28 | 28 days after randomization
  Ventilator free days to day 28 are defined as the number of days from the time of initiating unassisted breathing to day 28 after randomization, assuming survival for at least two consecutive calendar days after initiating unassisted breathing and continued unassisted breathing to day 28. If a patient returns to assisted breathing and subsequently achieves unassisted breathing to day 28, VFDs will be counted from the end of the last period of assisted breathing to day 28. A period of assisted breathing lasting less than 24 hours and for the purpose of a surgical procedure will not count against the VFD calculation. If a patient was receiving assisted breathing at day 27 or dies prior to day 28, VFDs will be zero.
Organ failure to day 5 | 5 days after randomization
  Organ failure is defined as present when the most abnormal vital signs or clinically available lab value meets the definition of clinically significant organ failure according to SOFA scores. Patients will be followed daily from randomization to day 5 for development of organ failures.
Mortality at day 28 | 28 days after randomization
  The occurrence of death in the ICU will be recorded until day 28.
Length of ICU-stay up to 28 days | 28 days after randomization
  The total number of days from admission to ICU discharge will be recorded until day 28
Physiological measures: Oxygenation | 28 days after randomization
  - Oxygenation Index on study days 1-5
Physiological measures: PaCO2 | 28 days after randomization
  - PaCO2 on study days 1-5
Physiological measures: pH | 28 days after randomization
  - Arterial pH on study days 1-5
Physiological measures: PEEP | 28 days after randomization
  - Level of PEEP (and static auto-PEEP in patients under controlled ventilation) on study days 1-5
Physiological measures: Plateau pressure | 28 days after randomization
  - Plateau pressure, static compliance of the respiratory system on study day 1-5
Physiological measures: Pneumothorax | 28 days after randomization
  - Development of pneumothorax through day 28
Physiological measures: Switch from controlled to pressure-support ventilation | 28 days after randomization
  - Time to switching from controlled to pressure-support ventilation through day 5
Physiological measures: Airway occlusion pressure | 28 days after randomization
  - Airway occlusion pressure at 0.1 s (P0.1), an index of respiratory drive, on the day the patient is switched to pressure-support ventilation if within 5 days since randomization
Hemodynamic measures | 28 days after randomization
  - Hemodynamic measures (mean arterial pressure, dose of infused norepinephrine or other vasopressor, serum lactate level) on study days 1-5
Physiological measures: Acute kidney injury | 28 days after randomization
  - KDIGO criteria for acute kidney injury 24 through day 5
Physiological measures: Supraventricular tachycardia | 28 days after randomization
  - Supraventricular tachycardia (SVT) or new onset atrial fibrillation through day 5
ICU-acquired delirium | 28 days after randomization
  The Confusion Assessment Method for the ICU (CAM-ICU, Appendix C )97 will be assessed daily from study entry to study day 28, death or ICU discharge, whichever comes first.
Biomarker measurements | from inclusion to 5 days
  Plasma samples will be collected from indwelling catheters (when available) at study entry and on days 1, 2, 3, 4, 5 in order to assemble a biological collection aimed at further investigating the effects of inhaled sedation with sevoflurane in patients with ARDS.
  The investigators will also collect whole blood samples at study entry and on day 2 for future studies of macrophage activation profiles and RNA and DNA studies.

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Not Required For This Country, France